CLINICAL TRIAL: NCT04189861
Title: The Role of Brain Wave Monitoring in Reducing the Incidence of Postoperative Cognitive Dysfunction
Brief Title: Use of Brain Wave Monitoring During Surgery to Reduce Postoperative Cognitive Dysfunction
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Myles D. Boone, MD MPH, Staff Physician, Anesthesiology, Dartmouth-Hitchcock Medical Center
Other Study IDs: D19171
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research study is being done to determine if indices derived from monitoring brain wave activity while under general anesthesia will predict the likelihood of post-operative cognitive dysfunction in patients over 60 years old.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) occurs in 30-40% of older adults after undergoing surgical procedures. POCD be subtle, such as a formerly avid reader unable to read for comprehension, to more overt, such as the inability to perform self-care. This deterioration in cognitive function leads to increased mortality, premature departure from the labor market and economic hardship. With 25 million people over the age of 60 undergoing surgical procedures annually in the United States and most of them living long into their 8th decade, prevention of POCD is an important public health issue.

The causal mechanism of POCD remains unclear, though older patients who receive general anesthesia are at increased risk relative to younger patients. While the association between age and POCD is not fully understood, several normal, age-related changes to brain anatomy and physiology may explain the increased susceptibility. These include decreased brain volume, notably in the prefrontal cortex, cortical thinning and altered neurotransmitter function. Taken together, these changes decrease the anesthetic requirements for older patients to achieve a similar anesthetic state and make them susceptible to overdosing of anesthetic agents. This is supported by studies using electroencephalography (EEG) to measure cerebral cortical activity which have demonstrated profound age-related differences for patients receiving general anesthesia. Older patients are more likely to develop burst suppression, an EEG pattern associated with an excessive anesthetic state. Currently, a major limitation in the field is the absence of studies that have used raw EEG data to examine the association between the dosing of anesthetic agents and POCD in older patients. Although prior studies have used EEG-derived depth of anesthesia indices to explore this association, these indices have been shown to be an unreliable measure of anesthetic state in older patients. Thus, the question of whether an excessive anesthetic state in this population causes POCD remains unanswered.

The investigators will recruit 100 adults over 60 years of age who undergo elective surgery under general anesthesia with EEG monitoring. A brief neurocognitive test battery will be conducted before surgery, 3-7 day post-surgery, and 3 months post-surgery to assess the association between EEG suppression and POCD.

In this study, the investigators hypothesize that the duration of EEG suppression is associated with POCD.

ELIGIBILITY:
Inclusion Criteria:

* 60-80 years of age who present for elective, non-cardiac surgical procedure requiring general anesthesia and an anticipated two-day or longer inpatient hospital stay
* English as the native and primary language
* Presence of an informant who has had weekly contact with the participant for at least the last year
* Participant is capable of providing written informed consent.

Exclusion Criteria:

* history of persistent and severe mental illness (e.g., schizophrenia, bipolar disorder)
* neurological disorder (e.g., Parkinson's disease, epilepsy, stroke)
* active substance use disorder as defined by the Diagnostic and Statistical Manual Diploma in Social Medicine(DSM-V)
* history of prior diagnosis of learning disability per the DSM-V
* estimated premorbid intellectual functioning below a scaled score of 70 based on the Test of Premorbid Functioning (TOPF)
* severe visual or hearing impairments that prevent the participant from undergoing the neurocognitive assessment.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60-80 years of age who present for elective, non-cardiac surgical procedure requiring general anesthesia and an anticipated two-day or longer inpatient hospital stay
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Postoperative Cognitive Decline | 3 months postoperatively
  The investigators will use a Composite Cognitive Change Score (between baseline and 3 months) to determine POCD

SECONDARY OUTCOMES:
Effective and Functional Connectivity | Day of surgery
  The investigators will use a multi-channel EEG (standard 10-20 montage) to assess changes to effective and functional connectivity during general anesethesia

OTHER OUTCOMES:
Postoperative Delirium | Postoperative days 2-7
  The investigators will use CAM-ICU to screen for postoperative delirium

CONTACTS AND LOCATIONS:
Overall Officials: M. Dustin Boone, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steinmetz J, Christensen KB, Lund T, Lohse N, Rasmussen LS; ISPOCD Group. Long-term consequences of postoperative cognitive dysfunction. Anesthesiology. 2009 Mar;110(3):548-55. doi: 10.1097/ALN.0b013e318195b569. PMID 19225398
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Deiner S, Westlake B, Dutton RP. Patterns of surgical care and complications in elderly adults. J Am Geriatr Soc. 2014 May;62(5):829-35. doi: 10.1111/jgs.12794. Epub 2014 Apr 14. PMID 24731176
- [Background] Peters R. Ageing and the brain. Postgrad Med J. 2006 Feb;82(964):84-8. doi: 10.1136/pgmj.2005.036665. PMID 16461469
- [Background] Morrison JH, Baxter MG. The ageing cortical synapse: hallmarks and implications for cognitive decline. Nat Rev Neurosci. 2012 Mar 7;13(4):240-50. doi: 10.1038/nrn3200. PMID 22395804
- [Background] Brown EN, Purdon PL. The aging brain and anesthesia. Curr Opin Anaesthesiol. 2013 Aug;26(4):414-9. doi: 10.1097/ACO.0b013e328362d183. PMID 23820102
- [Background] Purdon PL, Pavone KJ, Akeju O, Smith AC, Sampson AL, Lee J, Zhou DW, Solt K, Brown EN. The Ageing Brain: Age-dependent changes in the electroencephalogram during propofol and sevoflurane general anaesthesia. Br J Anaesth. 2015 Jul;115 Suppl 1(Suppl 1):i46-i57. doi: 10.1093/bja/aev213. PMID 26174300